CLINICAL TRIAL: NCT02053389
Title: Promoting Shared Decision Making in Prostate Cancer Through Decision Aids
Brief Title: Testing Decision Aids About Early Stage Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Angela Fagerlin, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: F021723 - 060077; P50CA101451-10 (NIH)
Record Dates: First submitted 2013-12-19; First posted 2014-02-03 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Prostatic Neoplasms
Keywords: Patient-Physician communication; Decision Support Techniques; Health Communication; Physician-Patient Relationship; Decision Making
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DVD Decision Aid (Experimental): Eligible participants receive the written decision aid ("Making the Choice: Deciding What to Do About Early Stage Prostate Cancer") AND the DVD decision aid ("Discussing the Choice: Talking with your Doctor about Early Stage Prostate Cancer"), which provides instruction and recommendations on how to participate in shared decision making with one's physician.
  Interventions: Behavioral: DVD Decision Aid
- Written Decision Aid (Active Comparator): Eligible participants receive the written decision aid ("Making the Choice: Deciding What to Do About Early Stage Prostate Cancer") alone.
  Interventions: Behavioral: Written decision aid

INTERVENTIONS:
Behavioral: DVD Decision Aid — The decision aid, "Discussing the Choice: Talking with your Doctor about Early Stage Prostate Cancer" is a DVD modeling patient communication strategies. The DVD includes vignettes with actors depicting patient-physician discussions of prostate cancer treatments. In these vignettes, the patient models communication strategies designed to facilitate patient activation.
  Arms: DVD Decision Aid
Behavioral: Written decision aid — A written decision aid entitled "Making the Choice: Deciding What to Do About Early Stage Prostate Cancer" that describes treatment options for early stage prostate cancer.
  Arms: Written Decision Aid

SUMMARY:
This is an educational intervention study testing the effects of decision aids in promoting patient participation in early stage prostate cancer treatment decision making. The purpose of this study is to compare patient-physician communication between patients who receive a DVD that models patient communication strategies vs. those who do not receive a DVD. All patients will also receive a written decision aid that describes treatment options for early stage prostate cancer. The Investigators hypothesize that the DVD will:

* increase patients' perceptions of the importance of their preferences to their decision making
* increase patients' perceptions of their intention to discuss their values and preferences with their urologists and radiation oncologists
* increase patients' actual engagement with their physician during the clinical encounter
* increase the concordance between patient decision making preferences and actual decision making outcomes
* increase long term satisfaction with decision on type of treatment selected
* increase patient satisfaction with their decision and the decision making process
* influence patient perception of his physician (e.g., trust) and of the diagnosis visit

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 years and older
* Scheduled for a prostate biopsy to test for prostate cancer
* Ability to read and answer survey questions in English

Exclusion Criteria:

* Previous diagnosis of prostate cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 564 (Actual)
Dates: Start 2010-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Self-efficacy for discussing preferences (intention) | Time 1 (baseline)
  14 item survey instrument
Self-efficacy for discussing preferences (intention) | Time 2 (post-intervention, an average of 3 days after Time 1 baseline)
  14 item survey instrument
Self-efficacy for discussing preferences (actual) | Time 3 (post-diagnosis, an average of 1 month after Time 1 baseline)
  14 item survey instrument

SECONDARY OUTCOMES:
Preference for shared decision making | Time 1 (baseline)
  1 item survey instrument
Preference for shared decision making | Time 2 (post-intervention, an average of 3 days after Time 1 baseline)
  1 item survey instrument
Prostate cancer related knowledge | Time 1 (baseline)
  10 item survey instrument
Prostate cancer related knowledge | Time 2 (post-intervention, an average of 3 days after Time 1 baseline)
  10 item survey instrument
Prostate cancer related knowledge | Time 3 (post-diagnosis, an average of 1 month after Time 1 baseline)
  12 item survey instrument
Prostate cancer related anxiety | Time 1 (baseline)
  6 item survey instrument
Prostate cancer related anxiety | Time 2 (post-intervention, an average of 3 days after Time 1 baseline)
  6 item survey instrument
Prostate cancer related anxiety | Time 3 (post-diagnosis, an average of 1 month after Time 1 baseline)
  6 item survey instrument
Prostate cancer related anxiety | Time 4 (6 months post diagnosis)
  7 item survey instrument
Treatment preference | Time 2 (post-intervention, an average of 3 days after Time 1 baseline)
  1 item survey instrument
Treatment decision | Time 3 (post-diagnosis, an average of 1 month after Time 1 baseline)
  2 item survey instrument
Treatment decision | Time 4 (6 months post diagnosis)
  2 item survey instrument
Decisional regret | Time 4 (6 months post diagnosis)
  5 item survey instrument
Preference for shared decision making | Time 3 (post-diagnosis, an average of 1 month after Time 1 baseline)
  1 item survey instrument
Preference for shared decision making | Time 4 (6 months post diagnosis)
  1 item survey instrument

CONTACTS AND LOCATIONS:
Overall Officials: Angela T Fagerlin, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Fridman I, Ubel PA, Kahn VC, Fagerlin A. Association of quantitative information and patient knowledge about prostate cancer outcomes. Health Psychol. 2022 Jul;41(7):484-491. doi: 10.1037/hea0001196. PMID 35727324